CLINICAL TRIAL: NCT06069193
Title: Effects of Physical Touch on Treatment Outcomes and Patient Perception in Individuals With Back and Neck Pain: an Experimental Study
Brief Title: Enhancing Treatment Outcomes: The Impact of Physical Touch in Back and Neck Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PainTouchOutcomes
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pain
Keywords: randomized controlled trial; placeboresponse; pain; doctor-patient interaction; treatment expectations
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two experimental groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants were not aware which experimental condition they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Touch Intervention (Experimental): This group receives professional touch techniques, such as procedural touch.
  Interventions: Behavioral: Touch Intervention
- Experimental: Control (Experimental): This group does not receive professional touch techniques and serves as the control for comparison.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Touch Intervention — The participants will be examined, with various areas in the neck and upper back being palpated. Subsequently, the exercises to be performed at home will be demonstrated by the experimenter. The experimenter will ensure correct execution by touching specific areas in the neck and upper back of the participants. Finally, the participants will be provided with a cream to be applied to the affected regions.
  Placebo cream:
  The participants receive an inert placebo cream, which is a standard basic cream infused with lemon oil, produced by a local pharmacy. Participants are informed that they are about to receive an effective analgesic cream.
  Placebo exercises:
  Participants are assigned a series of five core exercises, with an optional supplementary exercise available in case any of the core exercises proves ineffective for the participants. Participants are led to believe that these exercises are expected to have therapeutic effects.
  Arms: Experimental: Touch Intervention
Behavioral: Control — The participants will be examined, and they will be asked to describe as accurately as possible the regions where they experience pain. Subsequently, the experimenter will demonstrate the exercises to be performed at home. Finally, the participants will be provided with a cream to be applied to the affected regions.
  Placebo cream:
  The participants receive an inert placebo cream, which is a standard basic cream infused with lemon oil, produced by a local pharmacy. Participants are informed that they are about to receive an effective analgesic cream.
  Placebo exercises:
  Participants are assigned a series of five core exercises, with an optional supplementary exercise available in case any of the core exercises proves ineffective for the participants. Participants are led to believe that these exercises are expected to have therapeutic effects.
  Arms: Experimental: Control

SUMMARY:
In this study, we aim to investigate the impact of professional touch techniques on treatment expectations and adherence in German-speaking adults with current back or neck pain. Participants will engage in a 45-minute interaction, including structured components and physical touch interventions. We will assess treatment expectations, treatment effects, adherence, and participant motivation. Our study will provide insights into the role of touch in healthcare interactions and its influence on treatment outcomes.

DETAILED DESCRIPTION:
Research findings indicate that the interaction between healthcare professionals and patients can significantly influence both treatment expectations and their effectiveness. A compassionate, caring, and attentive doctor-patient interaction plays a crucial role in patient satisfaction and promotes accelerated recovery. Moreover, patient expectations are not solely shaped by interactions with healthcare providers but are also conceptualized through conditioning processes as one of the key mechanisms of the placebo effect. The effective performance of medical staff can further intensify patient expectations, contributing to an increased placebo response. While the effects of verbal communication on the placebo effect have been extensively studied, there is less research on the impact of nonverbal factors such as touch. Touch is a fundamental aspect of social interaction that can positively affect well-being and health. Touch is regarded as a mechanism for the positive health effects of social relationships and plays a significant role in bonding, communication, and reward. Physical touch can provide patients with a sense of presence and grounding, helping them feel seen, reassured, relaxed, and validated. In medical treatment, touch can enhance a sense of being taken seriously and cared for, thereby alleviating suffering and improving well-being. However, the full range of communicative potential in professional touch remains largely untapped, while a well-founded interdisciplinary synthesis is still lacking. For the planned study, we aim to recruit German-speaking adult participants who report current back or neck pain. Recruitment will be carried out through targeted outreach via various channels such as mailing lists, internet forums, and flyers. In an online experiment, we will initially assess baseline treatment expectations and current pain intensity. Subsequently, participants will be randomized into two experimental conditions. Participants will engage in a 45-minute interaction, comprising a structured opening, a brief interview, a standardized diagnostic examination, a detailed explanation of the pain relief cream, specific exercises, and a final farewell. Within the two experimental groups, physical interaction, specifically the application of professional touch techniques, in the form of procedural touch (serving diagnostic or therapeutic purposes), will be manipulated by aspiring pain specialists to examine its influence on various treatment parameters such as treatment expectations, treatment effects, treatment adherence, and participant motivation. Additionally, perceived empathy as well as warmth and competence of the treating person will be analyzed as relevant factors. Following the interaction, participants will be asked to perform specific exercises daily for one week and apply a placebo cream. Adherence to these medical and behavioral measures is a critical outcome criterion. At the end of the study, a systematic assessment of relevant behavioral parameters will be conducted to quantify potential changes in participants' behavior related to the interventions performed.

ELIGIBILITY:
Inclusion Criteria:

* Present complaints of back or neck pain
* Age of at least 18 years
* Proficiency in the German language
* Willingness to engage in daily short exercise routines

Exclusion Criteria:

* NRS <3 at baseline (0 = no pain and 10 = worst possible pain)
* Presence of contraindications for physical activity, such as severe disc diseases
* Presence of a severe medical condition
* Initiation of new pain treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity (Numerical Rating Scale (NRS)) | Pre-treatment (baseline); after the intervention (45 minutes after baseline); Post-treatment (1-week after baseline)
  Change in subjective pain intensity assessed using a numerical rating scales (NRS) ranging from 0 to 10, with higher values reflecting more pain intensity.
Change in treatment expectation (Generic Rating for Treatment Pre-Experiences, Treatment Expectations, and Treatment Effects, G-EEE) | Pre-treatment (baseline); after the intervention (45 minutes after baseline)
  Change from baseline in scores on the subscale for treatment expectations of the the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) Treatment expectations are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences and subscale for treatment expectations (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)
Treatment effects (Generic Rating for Treatment Pre-Experiences, Treatment Expectations, and Treatment Effects, G-EEE) | Post-treatment (1-week after baseline)]
  Treatment effects are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences and subscale for treatment expectations (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)

SECONDARY OUTCOMES:
Perceived physician empathy (The consultation and relational empathy (CARE)) | After the intervention (45 minutes after baseline)]
  This instrument, rated by patients, examines the quality of interpersonal interactions in healthcare encounters. It consists of ten items, each assessed on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree), with higher scores idicating reduced levels of empathy displayed by physicians.
Warmth and competence ratings of the practioner | After the intervention (45 minutes after baseline)
  Participant perceptions of warmth and competence of the practitioner are measured via the Warmth and Credibility Screener - German translation: 12 items assessing perceived warmth (6 items) and competence (6 items) on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater ratings of warmth and competence (Seewald & Rief, submitted for publication; English original by Fiske et al., 2002.)
Treatment adherence (Exercise Adherence Rating Scale (EARS)) | Post-treatment (1-week after baseline)
  The Exercise Adherence Rating Scale (EARS) is a self-administrated questionnaire designed to measure adherence to prescribed home-based exercises. The EARS consists of six items that measure adherence and 10 items related to reasons for nonadherence. The items were scored using a 5-point Likert scale ranging from 0 = completely agree to 4 = completely disagree with a possible summed score range from 0 to 64. Positively phrased items were reversed scored so that a higher overall adherence score indicated better adherence to exercise.
Adherence (Behavioral Measure) | Post-treatment (1-week after baseline)
  Self-report on the number of days participants have fully completed the prescribed exercises and properly applied the cream.

OTHER OUTCOMES:
Sociodemographic variables | Baseline
  Gender, age, education, employment, nationality, mother tongue etc.
Warmth and competence ratings of the respondent | After the intervention (45 minutes after baseline)
  Self-assessment of the subject's warmth and competence via the Warmth and Credibility Screener - German translation: 12 items assessing perceived warmth (6 items) and competence (6 items) on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater ratings of warmth and competence (Seewald & Rief, submitted for publication; English original by Fiske et al., 2002.)
Attitude towards social touch (Social Touch Questionnaire (STQ)) | Baseline
  The STQ assessed the individual attitude towards touch. It comprises 20 items that are to be answered on a 5-point Likert-scale from 0 (not at all) to 4 (extremely).
Anxiety (State-Trait Anxiety Inventory (STAI)) | Baseline
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 40-item self-administered questionnaire designed to assess both immediate state anxiety (reflecting current feelings at the moment) and long-term trait anxiety (reflecting general anxiety tendencies) with 20 items each. Participants rate their responses on a 4-point Likert scale, ranging from 1 (indicating "not at all" for state anxiety or "almost never" for trait anxiety) to 4 (indicating "very much so" for state anxiety or "almost always" for trait anxiety. According to the developer (Spielberger, 1983), scores of 20-39, 40-59, and 60-80 indicate low, moderate, and high anxiety, respectively.
Problems and Obstacles During the Intervention | Post-treatment (1-week after baseline)
  Problems with the execution of daily exercises were recorded in the online survey using an open response format.
Experiences with Physiotherapy | Post-treatment (1-week after baseline)
  The experience with physiotherapy is recorded on a 10-point scale from 0=never to 10=very frequent. High values represent a lot of experience with physiotherapy.
Parallel Treatments | Post-treatment (1-week after baseline)
  Treatments that were received during the participation period are selected in the survey (e.g., primary care treatment, orthopedic treatment). If a treatment is not listed, there is an option to specify it in an open field.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Dept. of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Germany
Locations (1):
- Germany Philipps University, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prichard C, Newcomb P. Benefit to Family Members of Delivering Hand Massage With Essential Oils to Critically Ill Patients. Am J Crit Care. 2015 Sep;24(5):446-9. doi: 10.4037/ajcc2015767. PMID 26330438
- [Background] Carter A, Sanderson H. Complementary therapy. The use of touch in nursing practice. Nurs Stand. 1995 Jan 11-17;9(16):31-5. doi: 10.7748/ns.9.16.31.s37. PMID 7888321
- [Background] Chang SO. The conceptual structure of physical touch in caring. J Adv Nurs. 2001 Mar;33(6):820-7. doi: 10.1046/j.1365-2648.2001.01721.x. PMID 11298220
- [Background] Cocksedge S, George B, Renwick S, Chew-Graham CA. Touch in primary care consultations: qualitative investigation of doctors' and patients' perceptions. Br J Gen Pract. 2013 Apr;63(609):e283-90. doi: 10.3399/bjgp13X665251. PMID 23540485
- [Background] Czerniak E, Biegon A, Ziv A, Karnieli-Miller O, Weiser M, Alon U, Citron A. Manipulating the Placebo Response in Experimental Pain by Altering Doctor's Performance Style. Front Psychol. 2016 Jun 30;7:874. doi: 10.3389/fpsyg.2016.00874. eCollection 2016. PMID 27445878
- [Background] Fiske ST, Cuddy AJ, Glick P, Xu J. A model of (often mixed) stereotype content: competence and warmth respectively follow from perceived status and competition. J Pers Soc Psychol. 2002 Jun;82(6):878-902. PMID 12051578
- [Background] Fuentes J, Armijo-Olivo S, Funabashi M, Miciak M, Dick B, Warren S, Rashiq S, Magee DJ, Gross DP. Enhanced therapeutic alliance modulates pain intensity and muscle pain sensitivity in patients with chronic low back pain: an experimental controlled study. Phys Ther. 2014 Apr;94(4):477-89. doi: 10.2522/ptj.20130118. Epub 2013 Dec 5. PMID 24309616
- [Background] Gallace A, Spence C. The science of interpersonal touch: an overview. Neurosci Biobehav Rev. 2010 Feb;34(2):246-59. doi: 10.1016/j.neubiorev.2008.10.004. Epub 2008 Oct 17. PMID 18992276
- [Background] Kaptchuk TJ. The placebo effect in alternative medicine: can the performance of a healing ritual have clinical significance? Ann Intern Med. 2002 Jun 4;136(11):817-25. doi: 10.7326/0003-4819-136-11-200206040-00011. PMID 12044130
- [Background] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493
- [Background] Kelley JM, Lembo AJ, Ablon JS, Villanueva JJ, Conboy LA, Levy R, Marci CD, Kerr CE, Kirsch I, Jacobson EE, Riess H, Kaptchuk TJ. Patient and practitioner influences on the placebo effect in irritable bowel syndrome. Psychosom Med. 2009 Sep;71(7):789-97. doi: 10.1097/PSY.0b013e3181acee12. Epub 2009 Aug 6. PMID 19661195
- [Background] Kelly MA, Nixon L, McClurg C, Scherpbier A, King N, Dornan T. Experience of Touch in Health Care: A Meta-Ethnography Across the Health Care Professions. Qual Health Res. 2018 Jan;28(2):200-212. doi: 10.1177/1049732317707726. Epub 2017 May 11. PMID 29235944
- [Background] Kim SS, Kaplowitz S, Johnston MV. The effects of physician empathy on patient satisfaction and compliance. Eval Health Prof. 2004 Sep;27(3):237-51. doi: 10.1177/0163278704267037. PMID 15312283
- [Background] Lapp HS, Croy I. Insights from the German Version of the Social Touch Questionnaire: How Attitude towards Social Touch relates to Symptoms of Social Anxiety. Neuroscience. 2021 Jun 1;464:133-142. doi: 10.1016/j.neuroscience.2020.07.012. Epub 2020 Jul 13. PMID 32673628
- [Background] Mercer SW, Maxwell M, Heaney D, Watt GC. The consultation and relational empathy (CARE) measure: development and preliminary validation and reliability of an empathy-based consultation process measure. Fam Pract. 2004 Dec;21(6):699-705. doi: 10.1093/fampra/cmh621. Epub 2004 Nov 4. PMID 15528286
- [Background] Neumann M, Wirtz M, Bollschweiler E, Warm M, Wolf J, Pfaff H. [Psychometric evaluation of the German version of the "Consultation and Relational Empathy" (CARE) measure at the example of cancer patients]. Psychother Psychosom Med Psychol. 2008 Jan;58(1):5-15. doi: 10.1055/s-2007-970791. Epub 2007 Apr 11. German. PMID 17429761
- [Background] Newman-Beinart NA, Norton S, Dowling D, Gavriloff D, Vari C, Weinman JA, Godfrey EL. The development and initial psychometric evaluation of a measure assessing adherence to prescribed exercise: the Exercise Adherence Rating Scale (EARS). Physiotherapy. 2017 Jun;103(2):180-185. doi: 10.1016/j.physio.2016.11.001. Epub 2016 Nov 9. PMID 27913064
- [Background] Olsson B, Olsson B, Tibblin G. Effect of patients' expectations on recovery from acute tonsillitis. Fam Pract. 1989 Sep;6(3):188-92. doi: 10.1093/fampra/6.3.188. PMID 2792618
- [Background] Schedlowski M, Enck P, Rief W, Bingel U. Neuro-Bio-Behavioral Mechanisms of Placebo and Nocebo Responses: Implications for Clinical Trials and Clinical Practice. Pharmacol Rev. 2015 Jul;67(3):697-730. doi: 10.1124/pr.114.009423. PMID 26126649
- [Background] Thomas KB. General practice consultations: is there any point in being positive? Br Med J (Clin Res Ed). 1987 May 9;294(6581):1200-2. doi: 10.1136/bmj.294.6581.1200. PMID 3109581
- [Background] Wearn A, Clouder L, Barradell S, Neve H. A qualitative research synthesis exploring professional touch in healthcare practice using the threshold concept framework. Adv Health Sci Educ Theory Pract. 2020 Aug;25(3):731-754. doi: 10.1007/s10459-019-09901-9. Epub 2019 Jul 16. PMID 31312926
- [Background] Wilhelm FH, Kochar AS, Roth WT, Gross JJ. Social anxiety and response to touch: incongruence between self-evaluative and physiological reactions. Biol Psychol. 2001 Dec;58(3):181-202. doi: 10.1016/s0301-0511(01)00113-2. PMID 11698114